CLINICAL TRIAL: NCT03624452
Title: The Effects of 8 Weeks of Remote Ischaemic Preconditioning Combined With Exercise Training on (Cerebro) Vascular Function.
Brief Title: Remote Ischaemic Preconditioning Combined With Exercise Training on Vascular Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Exericse&rIPC
Record Dates: First submitted 2018-07-18; First posted 2018-08-10 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Disease Risk
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rIPC and exercise training (Experimental): Those in the rIPC + exercise group will attend three 50 minute exercise sessions per week for 8 weeks at Liverpool John Moores University and 3 bouts of IPC per week at home at a time of their choice
  Interventions: Other: rIPC + Exercise
- rIPC only (Experimental): Those randomly allocated into the rIPC group will self administer 3 bouts of IPC per week at home at a time of their choice.
  Interventions: Other: rIPC only

INTERVENTIONS:
Other: rIPC + Exercise — The interventions consist of exercise training on a static bike three times per week and/or three bouts of rIPC per week for 8 weeks. A single bout of rIPC consists of cycles of upper arm cuff inflation for 5 minutes, followed by 5 minutes cuff deflation repeated 4 times.
  Arms: rIPC and exercise training
Other: rIPC only — Three bouts of rIPC per week for 8 weeks. A single bout of rIPC consists of cycles of upper arm cuff inflation for 5 minutes, followed by 5 minutes deflation repeated 4 times.
  Arms: rIPC only

SUMMARY:
Remote Ischaemic preconditioning' (RIPC) is defined as short controlled sequences of repeated inflation of a blood pressure cuff on the upper arm (to reduce blood flow) for 5 mins followed by recovery (cuff deflation so blood flows normally again). An intervention consisting of 4 cycles of 5 min of arm cuff inflation followed by deflation performed 3 times per week, spread over 8 weeks has been shown to improve blood vessel function in young individuals without any medical conditions. This is a simple and easily applicable intervention that could help the blood vessels capacity to deliver blood to an organ (e.g. heart or the muscle).It is currently unknown if RIPC combined with exercise training, provides stronger benefits to our blood vessels than RIPC alone. Therefore, the aim of this study is to investigate if combining RIPC with an 8 week exercise training programme improves blood vessel health more than 8 weeks of RIPC alone.

DETAILED DESCRIPTION:
A bout of ischaemia using a blood pressure cuff on the upper arm inflated to a pressure of 220 mm Hg for 5 mins followed by reperfusion (deflation of the cuff) is commonly known as remote ischaemic preconditioning (RIPC). Traditionally, RIPC refers to 5 minutes of inflation-5 minutes deflation repeated 4 times. Recent research has investigated the impact of repeated RIPC interventions on cardiovascular health. One previous repeated RIPC intervention, whereby RIPC was performed 3 times per week for eight weeks, identified that RIPC significantly enhanced conduit artery endothelial function and microvascular function.

Exercise training is crucial for a healthy lifestyle, with the World Health Organization recommending that adults aged 18-64 should do at least 150 minutes of moderate aerobic physical activity per week, or at least 75 minutes of vigorous intensity activity. Interestingly, the impact of exercise training on the vasculature is similar to that of repeated RIPC interventions, with reductions in arterial blood pressure, increased in blood flow and improvements in systemic vascular endothelial function. No study has examined if combining exercise and RIPC provides enhanced effects on the vasculature compared to exercise alone.

The aim of this study is to investigate whether combining 8 weeks of exercise and RIPC is more beneficial to systemic vascular function that exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent.
* Males and females 18 to 65 years.
* Body Mass Index >30g/m2 or waist circumference of ≥94cm (male), ≥80cm (female).
* Raised blood pressure systolic >130 or diastolic >85 mmHg or normal
* Diagnosed with high cholesterol by GP or normal

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Previous myocardial infarction, stroke (including TIA) or thrombosis
* Diagnosed with Congestive Heart failure
* Unable to enroll for the duration of the study
* Pregnancy or lactation period
* Smoking
* Any arm injury that will prevent application of the RIPC-intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-17 (Actual)

PRIMARY OUTCOMES:
Changes in peripheral vascular function | Peripheral vascular function will be assessed before the intervention, after 2 weeks of the intervention and after the end of the 8 week intervention.
  Flow mediated dilation will be used to assess endothelial-dependent vasodilation of the brachial artery.

SECONDARY OUTCOMES:
Detect changes in cerebrovascular function | Cerebrovascular function will be assessed before the intervention, after 2 weeks of the intervention and after the end of the 8 week intervention.
  Transcranial Doppler will be used to assess the cerebral blood flow response to changes in blood pressure, neural activity and breathing rate.
Response to an ischemia re-perfusion injury | Assessments will be performed before the intervention, after 2 weeks of the intervention and after the end of the 8 week intervention.
  Vascular response to an ischemia re-perfusion injury will be assessed in the upper arm using 15 minutes of cuff inflation to 200mmHg followed by 15 minutes of reperfusion. The ability of the brachial artery to vasodilate will be used as a marker of reperfusion injury.
Assessment of cardiorespiratory fitness | Cardiorespiratory fitness will be assessed before and after the 8 week intervention
  This will involve assessment of cardiorespiratory fitness using a maximal oxygen uptake test on a treadmill. Participants will be fitted with a heart rate monitor and face mask.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Sport and Exercise Science, Liverpool John Moores Unversity, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No